CLINICAL TRIAL: NCT04041635
Title: Reduction of Visual and Auditory Stimuli to Reduce Pain During Venipuncture in Premature Infants. A Randomized Controlled Trial.
Brief Title: Reduction of Visual and Auditory Stimuli to Reduce Pain During Venipuncture in Premature Infants.
Acronym: VENOPUNCIPREM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI-18-208
Record Dates: First submitted 2019-07-25; First posted 2019-08-01 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Premature; Pain, Procedural
Keywords: Pain; Premature; Visual stimuli; Auditory stimuli
MeSH Terms: conditions — Premature Birth; Pain, Procedural; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimuli Reduction (Experimental): This group will receive reduced visual and auditory stimuli in addition to usual care during venipuncture. Phototherapy goggles and earmuffs will be placed 3 minutes before the venipuncture (leaving the patient in resting state after the manipulation) and will be maintained during the procedure. Monitor alarms and devices will be silenced and will remain silenced and noise in the unit will be minimized during the procedure.
  Interventions: Procedure: Stimuli reduction
- Usual Care (Active Comparator): Babies in the control group will receive physical contention with administration of sucrose two minutes before carrying out the venipuncture procedure (usual care). Venipuncture will be performed with 22G extraction needles, or peripheric venous catheter. During the puncture the eyes will not be covered, and monitor alarms and devices be not be silenced.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Stimuli reduction — Phototherapy goggles and earmuffs will be placed 3 minutes before the venipuncture (leaving the patient in resting state after the manipulation) and will be maintained during the procedure. Monitor alarms and devices will be silenced and will remain silenced and noise in the unit will be minimized during the procedure.
  Arms: Stimuli Reduction
Procedure: Usual care — Babies in the control group will receive physical contention with administration of sucrose two minutes before carrying out the venipuncture procedure (usual care). Venipuncture will be performed with 22G extraction needles, or peripheric venous catheter. During the puncture the eyes will not be covered, and monitor alarms and devices be not be silenced.
  Arms: Usual Care

SUMMARY:
The aim of the study is: To evaluate the efficacy of the reduction of visual and auditory stimuli on pain during venipuncture in premature newborns of 32-36 weeks of gestation.

DETAILED DESCRIPTION:
Background: The evidence for the efficacy of reducing sensory stimulation and its effect on pain in minor procedures has not been studied in depth. There are no studies that evaluate the reduction of visual and auditory stimuli in a combined way.

Impact: It is easy to incorporate the reduction of visual and auditory stimuli into nursing practice.

Aims: To evaluate the efficacy of the reduction of visual and auditory stimuli on pain during venipuncture in premature newborns of 32-36 weeks of gestation.

Design: Open, randomized, non-blind parallel clinical trial. Methods: Study to take place at the neonatal intensive care unit at the Germans Trias i Pujol University Hospital in 2019-2021. 56 recently born babies between 32 and 36 weeks of gestation will participate. The dependent variable is level of pain determined using the Premature Infant Pain Profile (PIPP). The intervention will be assigned randomly using the random.org software. Data analysis will be carried out using the IBM SPSS v.25 software assuming a level of significance of 5%.

The results of this study could have a direct impact on clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies born between 32 and 36 weeks of gestation (both included).
* Haemodynamically stable.
* Require venipuncture and whose.
* Parents or legal guardians have signed informed consent forms.

Exclusion Criteria:

* Gestational age inferior to 32 weeks.
* Treated with intravenous or oral analgesics, sedatives or relaxants.
* Critical status or haemodynamically unstable.
* Requiring invasive mechanical ventilation.

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Premature Infant Pain Profile (PIPP) score | From baseline Pain determination at (just before venipuncture) to 30 seconds after venipuncture
  Calculation of pain response using a validated instrument (Premature Infant Pain Profile-PIPP). It varies from "0" (no pain to 21 (maximum pain response)

SECONDARY OUTCOMES:
Change in heart rate | From baseline Pain determination at (just before venipuncture) to 30 seconds after venipuncture
  Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bonjorn-Juarez, RN, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Bonjorn Juarez M, Manrique Pons M, Grau Alcon L, Martinez-Momblan MA, Alonso-Fernandez S. Reduction of visual and auditory stimuli to reduce pain during venipuncture in premature infants. Study protocol for a randomized controlled trial. J Adv Nurs. 2020 Apr;76(4):1077-1081. doi: 10.1111/jan.14300. Epub 2020 Jan 10. PMID 31865625